CLINICAL TRIAL: NCT02648815
Title: Management of Moderate and Severe Forms of Acute Pancreatitis
Brief Title: Management of Pancreatitis: the Role of Supportive and Drainage Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Clinical Center Tuzla (Other)
Responsible Party: Principal Investigator, Enver Zerem, Professor of medicine, University Clinical Center Tuzla
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UClinicalCenterTuzla; 04-09/2-93/15 (Other: University Clinical Center Tuzla)
Record Dates: First submitted 2015-12-31; First posted 2016-01-07 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatitis
Keywords: Necrotizing pancreatitis; Sepsis; Infection; Drainage
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing; Sepsis; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous catheter drainage group (Active Comparator): Percutaneous catheter drainage (PCD) of necrotic tissue and pathological collections formed during acute pancreatitis
  Interventions: Procedure: Percutaneous catheter drainage
- Abdominal paracentesis evacuation group (Active Comparator): Abdominal paracentesis drainage (APD) of peritoneal fluid during acute pancreatitis
  Interventions: Procedure: Abdominal paracentesis evacuation

INTERVENTIONS:
Procedure: Percutaneous catheter drainage — Depending on the operator experience, tandem trocar technique or Seldinger technique can be used. If the Seldinger technique is used, then the catheter tract should be sequentially dilated over a guidewire. Access routes that avoid crossing the bowel and other intervening organs, or major mesenteric, peripancreatic, or retroperitoneal blood vessels are selected to minimize the risk of bacterial contamination and hemorrhage. Successful percutaneous treatment of necrotic collections of the pancreas depends on several important factors. Catheters often need to remain in place for several weeks and sometimes months; hence, close follow-up is required.
  Arms: Percutaneous catheter drainage group
Procedure: Abdominal paracentesis evacuation — Evacuation of peritoneal ascitic fluid using percutaneous catheters
  Arms: Abdominal paracentesis evacuation group

SUMMARY:
This study aims to investigate the natural clinical course, diagnostic possibilities and treatment modalities in moderately severe (MSAP) and severe acute pancreatitis (SAP). The management of severe acute pancreatitis varies with the severity and depends on the type of complication that requires treatment. Although no universally accepted treatment algorithm exists, the step-up approach using close monitoring, percutaneous or endoscopic drainage, followed by minimally invasive video-assisted retroperitoneal debridement has demonstrated to produce superior outcomes to traditional open necrosectomy and may be considered as the reference standard intervention for this disorder.

DETAILED DESCRIPTION:
Despite overall reduced mortality in the last decade, MSAP and SAP are devastating diseases associated with mortality ranging from less than 10% to as high as 85%, according to various studies. The management of SAP is complicated because of the limited understanding of the pathogenesis and multi-causality of the disease, uncertainties in outcome prediction and few effective treatment modalities. Generally, sterile necrosis can be managed conservatively in the majority of cases with a low mortality rate (12%). However, infection of pancreatic necrosis can be observed in 25%-70% of patients with necrotizing disease; it is generally accepted that the infected non-vital tissue should be removed to control the sepsis. Laparotomy and immediate debridement of the infected necrotic tissue have been the gold standard treatment for decades. However, several reports have shown that early surgical intervention for pancreatic necrosis could result in a worse prognosis compared to cases where surgery is delayed or avoided. Therefore, several groups worldwide have developed new, minimally invasive approaches for managing infected necrotizing pancreatitis. The applicability of these techniques depends on the availability of specialized expertise and a multidisciplinary team dedicated to the management of SAP and its complications.

ELIGIBILITY:
Inclusion Criteria:

1. fluid collections within two weeks of disease onset;
2. single- or multi-organ failure;
3. CTSI > = 7 (initial CT performed within 7 days after the onset of disease.); and (4) acute physiology and chronic health evaluation (APACHE) II score > = 8.

Exclusion Criteria:

1. patients without APD interventions;
2. patients who underwent necrosectomy directly after APD without PCD as a bridge therapy;
3. previous percutaneous drainage or surgical necrosectomy during the episode of pancreatitis;
4. previous exploratory laparotomy for acute abdomen and intraoperative diagnosis of AP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants converted to more aggressive treatment | An average of 1 year

SECONDARY OUTCOMES:
Proportion of patients requiring PCD after initial APD | An average of 1 year
Morbidity and mortality in patients requiring PCD | An average of 1 year
Number of PCD interventions required | An average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Enver Zerem, MD.PhD, Principal Investigator — University Clinical Center Tuzla

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zerem E. Treatment of severe acute pancreatitis and its complications. World J Gastroenterol. 2014 Oct 14;20(38):13879-92. doi: 10.3748/wjg.v20.i38.13879. PMID 25320523
- [Result] Zerem E, Imamovic G, Susic A, Haracic B. Step-up approach to infected necrotising pancreatitis: a 20-year experience of percutaneous drainage in a single centre. Dig Liver Dis. 2011 Jun;43(6):478-83. doi: 10.1016/j.dld.2011.02.020. Epub 2011 Apr 8. PMID 21478061
- [Result] Zerem E, Imamovic G, Omerovic S, Imsirovic B. Randomized controlled trial on sterile fluid collections management in acute pancreatitis: should they be removed? Surg Endosc. 2009 Dec;23(12):2770-7. doi: 10.1007/s00464-009-0487-2. Epub 2009 May 15. PMID 19444515